CLINICAL TRIAL: NCT03114930
Title: Study of the Prevalence of Complications Occurring in the Mother-newborn Couple During the First Month After Returning Home, Since the Introduction of Standard Outpatients (According to HAS 2014 Recommendations) at the Amiens-Picardie University Hospital
Acronym: COMPLISTAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI2015_843_0023
Record Dates: First submitted 2017-04-04; First posted 2017-04-14 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Mother-Child Relations; Maternity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard output (Other)
  Interventions: Other: To study the absence of increased complications and events occurring in the "mother-newborn"
- Non standard output (Other)
  Interventions: Other: To study the absence of increased complications and events occurring in the "mother-newborn"

INTERVENTIONS:
Other: To study the absence of increased complications and events occurring in the "mother-newborn" — To study the absence of increased complications and events occurring in the "mother-newborn" couple who made a "standard" exit compared to the "mother-newborn" couples who had benefited from an extra day of " Hospitalization in maternity.

SUMMARY:
Prior to the HAS recommendations of March 2014, the "mother - newborn" couple was discharged from the maternity home at 4 days after delivery by AVB and 5 days after caesarean section.

The stay in maternity allowed a follow-up of the newborn whose weight gain and the occurrence of a jaundice; And monitoring of the mother whose milky ascent and psychological feelings.

In March 2014, the HAS published new recommendations on maternity leave arrangements for the "mother - newborn" couple, the organization of postpartum follow - up for the mother and pediatric follow - up for the newborn. The HAS then defines so-called "optimal" conditions for so-called "standard" outputs, with 9 criteria to respect respectively for the mother and the newborn.

If the mother-to-newborn couple respects these so-called optimal conditions and is eligible according to the respective criteria, the latter leaves at home after 72 hours and before 96 hours for an AVB and after 96 completed hours and Before 120 hours for caesarean delivery.

As no pediatric discharge was done in the afternoons at the maternity hospital of Amiens, an arbitrary choice was made to allow a "standard" release to the "mother-newborn" couple only if the child was born between 00H00 and 11H59 so that his clinical examination of exit is carried out at 72 hours of the birth as recommended by the recommendations of the HAS.

These recommendations being recent (2014), no study has studied the impact and consequences on the triad "father / mother-newborn" of these exits including the occurrence of possible complications or events: re-hospitalizations again The early termination of breastfeeding, and whether the follow-up procedures advocated by the HAS are being followed.

ELIGIBILITY:
Inclusion Criteria:

* Be taken care of in the Maternity Department of the Amiens-Picardie University Hospital.
* Parents' agreement
* Mother and Newborn who meet the eligibility criteria of the HAS for a "standard" exit.

Mother :

* 1. Absence of a situation of psychological, social vulnerability, behaviors of addiction and severe dependencies
* 2. Adequate family and / or social support
* 3. Absence of chronic ill-balanced pathology
* 4. Absence of complications or pathologies requiring observation or continuous medical treatment
* 5. Absence of haemorrhage of the delivery, this one was checked and treated (if necessary)
* 6. Absence of active infection or signs of infection
* 7. Absence of thromboembolic signs
* 8. Controlled Pain
* 9. Satisfactory mother-child interactions

Child:

* 1. Newborn at term ≥ 37 weeks of amenorrhea, singleton and eutroph
* 2. Normal clinical examination performed imperatively 48 hours after birth and before discharge
* 3. Axillary temperature between 36 and 37 ° C or central between 36.5 and 37.5 ° C
* 4. Established feeding (if breastfeeding: observation of at least 2 feeds ensuring effective transfer of colostrum / milk recognized by the mother), urination and spontaneous stool emissions, established transit
* 5. Weight loss <8% of birth weight
* 6. Absence of jaundice requiring phototherapy according to the therapeutic indication curve and measurement of transcutaneous and / or blood bilirubin at the output referred to the nomogram (low risk and low intermediate risk only)
* 7. Lack of clinical or paraclinical evidence for infection; If risk factors of infection: recovered and negative biological and bacteriological samples
* 8. Planned neonatal screening and traceability
* 9. Post-partum follow-up after the organized event: an appointment with a referral professional within 48 hours following the exit or even in the week

Exclusion Criteria:

* Patient not speaking French
* Patient who does not meet the HAS criteria: newborn or ineligible mother (minor mother, non-singleton birth)
* Assumption in another department than the Maternity department of the CHU Amiens-Picardie.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
The occurrence of complications in the first month of life in the "mother-newborn" couple. | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens Picardie, Amiens, Picardie, France